CLINICAL TRIAL: NCT07302646
Title: Comparison of Iodinated Contrast Media Injection Protocols With Reduced Flow Rates and Volumes on Image Quality in Diagnostic Cerebral Angiography for the Evaluation of Unruptured Intracranial Aneurysms: Towards a Standardization of Practices
Brief Title: Optimizing Reduced-Flow, Low-Volume Contrast Protocols for Cerebral Angiography in Unruptured Aneurysms
Acronym: OPIAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9882; 2025-524884-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Interventional Neuroradiology
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard (Reference) (Active Comparator): A control group following the current standard protocol used in Strasbourg."
  Interventions: Radiation: Standard (Reference)
- Reduced volume - standard flow rate (Experimental): Experimental group evaluating reduction in injection volume
  Interventions: Radiation: Reduced volume - standard flow rate
- Standard volume - Reduced flow rate (Experimental): Experimental group evaluating reduction in flow rate
  Interventions: Radiation: Standard volume - Reduced flow rate
- Reduced volume and flow rate (Experimental): Experimental group evaluating reduction in injection volumes and flow rate
  Interventions: Radiation: Reduced volume and flow rate

INTERVENTIONS:
Radiation: Standard (Reference) — Selection visit (D-40 to D-7): Patient information on cerebral angiography (standard consultation) and study objectives. Delivery of the information document and reflection period. Verification of eligibility criteria.
  Inclusion visit (D0): Review of study objectives and Q&A. Final verification of eligibility criteria. Obtaining of free and informed consent. Randomisation and assignment to an injection protocol.
  Angiography performed according to standard practice, with image acquisition using the assigned injection protocol. Assessment of patient discomfort (EVS) and satisfaction (SAPS).
  Data collection: ICM volume injected/consumed, radiation dose, and examination duration.
  Image handling: Archiving and pseudonymisation of images for later analysis. End of participation: Patient participation ends after this visit.
  Arms: Standard (Reference)
Radiation: Reduced volume - standard flow rate — Selection visit (D-40 to D-7): Patient information on cerebral angiography (standard consultation) and study objectives. Delivery of the information document and reflection period. Verification of eligibility criteria.
  Inclusion visit (D0): Review of study objectives and Q&A. Final verification of eligibility criteria. Obtaining of free and informed consent. Randomisation and assignment to an injection protocol.
  Angiography performed according to standard practice, with image acquisition using the assigned injection protocol. Assessment of patient discomfort (EVS) and satisfaction (SAPS).
  Data collection: ICM volume injected/consumed, radiation dose, and examination duration.
  Image handling: Archiving and pseudonymisation of images for later analysis. End of participation: Patient participation ends after this visit.
  Arms: Reduced volume - standard flow rate
Radiation: Standard volume - Reduced flow rate — Selection visit (D-40 to D-7): Patient information on cerebral angiography (standard consultation) and study objectives. Delivery of the information document and reflection period. Verification of eligibility criteria.
  Inclusion visit (D0): Review of study objectives and Q&A. Final verification of eligibility criteria. Obtaining of free and informed consent. Randomisation and assignment to an injection protocol.
  Angiography performed according to standard practice, with image acquisition using the assigned injection protocol. Assessment of patient discomfort (EVS) and satisfaction (SAPS).
  Data collection: ICM volume injected/consumed, radiation dose, and examination duration.
  Image handling: Archiving and pseudonymisation of images for later analysis. End of participation: Patient participation ends after this visit.
  Arms: Standard volume - Reduced flow rate
Radiation: Reduced volume and flow rate — Selection visit (D-40 to D-7): Patient information on cerebral angiography (standard consultation) and study objectives. Delivery of the information document and reflection period. Verification of eligibility criteria.
  Inclusion visit (D0): Review of study objectives and Q&A. Final verification of eligibility criteria. Obtaining of free and informed consent. Randomisation and assignment to an injection protocol.
  Angiography performed according to standard practice, with image acquisition using the assigned injection protocol. Assessment of patient discomfort (EVS) and satisfaction (SAPS).
  Data collection: ICM volume injected/consumed, radiation dose, and examination duration.
  Image handling: Archiving and pseudonymisation of images for later analysis. End of participation: Patient participation ends after this visit.
  Arms: Reduced volume and flow rate

SUMMARY:
Over the past two decades, interventional neuroradiology (INR) has seen significant advances in terms of safety and radiation protection. However, the management of iodinated contrast media (ICM) administered to the patients remains problematic. There is currently no reference for applying the ALADA (As Low As Diagnostically Acceptable) principle to ICM. In this context, optimising injection parameters seems essential to limit patient risks while maintaining sufficient diagnostic quality. To achieve this, it is necessary to work on a standardised procedure: the most frequently performed being diagnostic cerebral angiography for initial assessment or follow-up of intracranial aneurysms (IA). The aim of this project is to demonstrate that the use of injection protocols with reduced flow rates and volumes would enable non-inferior results compared to the empirical protocol (used in our department) in terms of image quality for the assessment of ICA, while improving examination comfort for patients.

A Randomised controlled non-inferiority study involving a four-arm factorial design to evaluate the impact of different ICM injection strategies in diagnostic cerebral angiography. Four groups will be compared: three experimental groups evaluating reductions in injection volumes and/or flow rates, and a control group following the standard protocol currently used in Strasbourg University Hospitals. Each subject will be randomly assigned to a group, and all images will be acquired using the same protocol. By following the standard care pathway and implementing safety procedures to ensure diagnostic quality, patients will not undergo any changes to their usual care and will not run any increased risk of diagnostic error.

ELIGIBILITY:
Inclusion Criteria:

Adult participant at the time of consent (age between 18 and 80 years old);

Scheduled diagnostic cerebral angiography as part of routine care:

* Initial assessment of the IA (suspected or detected in non-invasive imaging);
* Follow-up of one or more IAs (treated or untreated);
* Conscious and oriented participant, able to undergo the procedure under simple local anaesthesia;
* Participant able to understand the objectives of the research and provide a dated, signed informed consent form;
* Participant able to answer oral or written questions (French-speaking or understanding French);
* For women of childbearing potential: negative serum β-HCG test at the inclusion visit;
* Participant covered by a social security health insurance plan.

Exclusion Criteria:

* Emergency cerebral angiography;
* Participants with other neurovascular conditions (AVM, AVF, etc.) in addition to an IA;
* Participants with any contraindication to the use of ICM;
* Pregnancy or breastfeeding;
* Participants whose physical or psychological condition requires sedation or general anaesthesia for the procedure;
* Participants with communication or cognitive disorders; Incapable participants (subject to legal protection measures: curatorship, guardianship, judicial protection, future protection mandate, family authorization).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Ratio of exploitable 2D and 3D images | 1 day
  Ratio of exploitable 2D and 3D images, assessed by radiographers, obtained with each injection protocol (reduced flow rates/standard volumes; reduced volumes/standard flow rates; reduced flow rates and volumes), compared to the standard/empirical protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Imagerie Interventionnelle Vasculaire Hôpitaux Universitaires de Strasbourg 1, place de l'Hôpital, 67 091 STRASBOURG Cedex, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided